CLINICAL TRIAL: NCT02313493
Title: Improving Mental Health in First Time Parents - A Randomized Controlled Pilot Study
Brief Title: Efficacy and Feasibility of Baby Triple P - a Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Lukka Popp, M.Sc., Ruhr University of Bochum
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RCT-Baby Triple P
Record Dates: First submitted 2014-12-07; First posted 2014-12-10 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Mental Disorders During Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baby Triple P parent training group (Experimental): The 8- session program delivered in four group sessions before birth and four telephone sessions after birth is developed for parents at the transition to parenthood or with a baby (up to 12 months of age).
  Interventions: Behavioral: Baby Triple P
- Care as usual control group (No Intervention)

INTERVENTIONS:
Behavioral: Baby Triple P
  Arms: Baby Triple P parent training group

SUMMARY:
In the present pilot study the feasibility and efficacy of Baby Triple P- an antenatal parent training- are investigated. Healthy becoming first time parents were randomly allocated to either the Baby Triple P parent-training group or a care as usual control group. It is expected that 78 couples of becoming first time parents are recruited. It is hypothesized that parents and their infants in the parent training group will show significantly less psychopathology / regulation problems and better partnership quality than participants in the control condition.

DETAILED DESCRIPTION:
In this pilot study, the efficacy and feasibility of the Baby Triple P parenting training is investigated in a pilot study using a randomized controlled trial. According to the efficacy of the parenting training, it is expected that parents in the training condition show higher scores on mental health scales (BSI-18) and quality of Partnership (PFB). Furthermore, it is expected that infants whose parents has taken part in the parenting training have lower severity ratings of regulatory disorders assessed with the Baby-DIPS diagnostic interview than infants of parents in the care as usual control condition.

ELIGIBILITY:
Inclusion Criteria:

* Becoming first time parent
* Participants have a basic level of German literacy which allows them to understand the Baby Triple P materials
* Unborn Baby is developing well and does not have a pre-diagnosed medical condition

Exclusion Criteria:

* Baby has a disability or pre-diagnosed medical condition.
* The parents are intellectually disabled

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-07 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Number of symptoms on the BSI 18 and the PFB-K | Before birth (T1), two months after birth (T2)
  The BSI 18 assessment gathers patient-reported data to help measure psychological distress and psychiatric disorders. The relationship questionnaire (PFB-K) assess partnership satisfaction.
Severity rating (0-8) of regulatory problems in infants | six months after birth (T3)
  Regulatory difficulties in crying, sleeping and feeding behavior in infants are assessed with a diagnostic interview (Baby-DIPS). The severity rating ranges from 0-8 (> 4 indicates a clinical referred disorder).

SECONDARY OUTCOMES:
Quality of parenting | Two months after birth (T2), six month after birth (T3)
  Parent-related behavior and cognitions are assessed with the Parenting Sense of Competence Scale (PSOC; T2,T3) with both parents and the Postpartum Bonding Questionnaire (PBQ;T2) only with mothers. Additionally, explorative questionnaires assess program specific parenting skills and educational elements as the number of soothing strategies the parents apply or the knowledge about an infants' development (T2, T3).
Number of symptoms on the EPDS, DASS-21 and the OSS-3 | Two months after birth (T2)
  The Edinburgh Postnatal Depression Scale (EPDS, T2) is a rating scale for measuring the severity of postnatal depression symptoms. The Depression Anxiety Stress Scales (DASS-21) assess symptoms of depressions, anxiety and stress. The Oslo Social Support Scale (OSS-3) measures the subjective amount of social support the parents get.

REFERENCES:
- [Derived] Popp L, Fuths S, Schneider S. The Relevance of Infant Outcome Measures: A Pilot-RCT Comparing Baby Triple P Positive Parenting Program With Care as Usual. Front Psychol. 2019 Oct 29;10:2425. doi: 10.3389/fpsyg.2019.02425. eCollection 2019. PMID 31736826
- [Derived] Popp L, Schneider S. Attention placebo control in randomized controlled trials of psychosocial interventions: theory and practice. Trials. 2015 Apr 11;16:150. doi: 10.1186/s13063-015-0679-0. PMID 25872619